CLINICAL TRIAL: NCT07096544
Title: CALM Study: Cardiomems Assisted Lvad Management
Acronym: CALM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 025-422
Record Dates: First submitted 2025-07-22; First posted 2025-07-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group: CardioMEMS Device (Experimental): For patients randomized to the intervention group, the CardioMEMS device will be implanted during a right heart catheterization procedure. The device will be positioned in the pulmonary artery and calibrated using a Swan-Ganz catheter. After implantation, PAP measurements will be taken daily using the home monitoring system provided to the patient. These readings will be transmitted wirelessly to the clinical team, who will review the data at least once per week. Adjustments to the patient's medical therapy and LVAD speed settings will be made based on the hemodynamic data provided by the CardioMEMS device.
  Interventions: Device: CardioMEMS Device
- Control Group: Standard of Care Monitoring (No Intervention): Patients in the control group will be monitored according to standard of care, which includes periodic evaluations of echocardiographic parameters (e.g., left ventricular size and function, aortic and mitral valve function, and right ventricular function), clinical assessments (e.g., NYHA classification, medication review, and physical examination), quality of life assessments using the Kansas City Cardiomyopathy Questionnaire (KCCQ), functional status evaluations with a six-minute walk test, and monitoring for adverse events such as heart failure-related hospitalizations, reoperations, and device-related complications.

INTERVENTIONS:
Device: CardioMEMS Device — The CardioMEMS device will be implanted during a right heart catheterization procedure. The device will be positioned in the pulmonary artery and calibrated using a Swan-Ganz catheter. After implantation, PAP measurements will be taken daily using the home monitoring system provided to the patient. These readings will be transmitted wirelessly to the clinical team, who will review the data at least once per week. Adjustments to the patient's medical therapy and LVAD speed settings will be made based on the hemodynamic data provided by the CardioMEMS device.
  Arms: Intervention Group: CardioMEMS Device

SUMMARY:
This prospective, open label, randomized, single-center pilot clinical trial will determine if the rate of heart failure related (HFR) hospitalizations is less in LVAD patients whose PAP is monitored with the CardioMEMS device vs the control patients receiving standard of care treatment.

DETAILED DESCRIPTION:
This prospective, open label, randomized, single-center pilot clinical trial will determine if the rate of heart failure related (HFR) hospitalizations is less in LVAD patients whose PAP is monitored with the CardioMEMS device vs the control patients receiving standard of care treatment.

Secondary objectives:

* Number of emergency department visits
* Days alive outside the hospital
* Rate of all cause rehospitalizations
* Change in NYHA functional class
* Impact on quality of life as determined by utilizing the Kansas City Cardiomyopathy Questionnaire (KCCQ).
* Impact on functional status as determined by a six-minute walk test
* Rate of LVAD and CardioMEMS device malfunctions
* Change in baseline pulmonary pressures
* Rate and method of mortality

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85
* Status post HeartMate III Left Ventricular Assist Device Implantation
* Normally functioning left ventricular assist device as determined by device parameters
* Stable and ready to be discharged home
* 18 years of age or older at the time of left ventricular device implantation
* The patient provides written informed consent before starting any component of this clinical investigation

Exclusion Criteria:

* Current/ongoing fevers or constitutional symptoms
* Bilirubin greater than 2.5µmol/L, shock liver, or biopsy-proven liver cirrhosis
* Requiring dialysis or declared end stage renal disease
* Inability to complete written informed consent or a quality-of-life questionnaire
* Known active malignancy
* History of recurrent (> 1) pulmonary embolism or deep vein thrombosis
* Unable to tolerate a right heart catheterization
* Major cardiovascular event (e.g., myocardial infarction, stroke) within 2 months of CardioMEMS implant
* Glomerular Filtration Rate (GFR) <25 ml/min who are non-responsive to diuretic therapy
* Patients likely to undergo heart transplantation within 6 months of Screening Visit
* Congenital heart disease or mechanical right heart valve(s)
* Known coagulation disorders
* Hypersensitivity or allergy to aspirin, and/or clopidogrel
* Pregnant or considering pregnancy
* Required RV assist device and has severe right heart failure post LVAD implantation

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Heart failure related (HFR) hospitalizations | Through study completion, an average of 1 year
  Rate of heart failure related (HFR) hospitalizations in LVAD patients whose PAP is monitored with the CardioMEMS device vs the control patients receiving standard of care treatment.

SECONDARY OUTCOMES:
Emergency Visits | Through study completion, an average of 1 year
  Number of emergency department visits
Days alive outside the hospital | Through study completion, an average of 1 year
  Days alive outside the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White The Heart Hospital - Plano, Plano, Texas, United States

REFERENCES:
- [Background] Leff JP. Assessment of drugs in schizophrenia. Br J Clin Pharmacol. 1976 Feb;3(1 Suppl 1):75-8. doi: 10.1111/j.1365-2125.1976.tb03718.x. No abstract available. PMID 9960
- [Background] Hamar J, Ligeti L, Kovach AG. Intestinal O2 consumption under low flow conditions in anaesthetized cats. Adv Exp Med Biol. 1977 Jul 4-7;94:573-8. doi: 10.1007/978-1-4684-8890-6_77. No abstract available. PMID 26184
- [Background] Im WB, Christensen HN, Sportes B. Amino acid stimulation of ATP cleavage by two Ehrlich cell membrane preparations in the presence of ouabain. Biochim Biophys Acta. 1976 Jun 17;436(2):424-37. doi: 10.1016/0005-2736(76)90205-4. PMID 6067
- [Background] Collins MW, French MR, Hirom PC, Idle JR, Bassir O, Williams RT. The conjugation of benzoic acid in the African bat, Epomops franqueti. Comp Biochem Physiol C Comp Pharmacol. 1977;56(2):103-4. doi: 10.1016/0306-4492(77)90021-1. No abstract available. PMID 15767